CLINICAL TRIAL: NCT02197429
Title: Acupuncture for the Treatment of Vulvodynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schlaeger, Judith M., CNM, LAc, PhD (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-10-01
Record Dates: First submitted 2014-07-14; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Vulvodynia; Vulvar Vestibulitis; Pain; Dyspareunia; Female Sexual Dysfunction Due to Physical Condition
Keywords: Vulvodynia; Acupuncture; Provoked Vestibulodynia; Vulvar Vestibulitis; Vulvar Pain; Dyspareunia; Female Sexual Function
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis; Pain; Dyspareunia | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture
  Interventions: Other: Acupuncture
- Wait-list Control (No Intervention): Wait-list Control

INTERVENTIONS:
Other: Acupuncture
  Arms: Acupuncture

SUMMARY:
A randomized controlled pilot study was conducted to evaluate the effect of an acupuncture protocol for the treatment of vulvodynia.

Hypotheses:

1. Acupuncture reduces vulvar pain and dyspareunia in women with vulvodynia.
2. Acupuncture increases sexual function in women with vulvodynia.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with either generalized vulvodynia, localized vestibulodynia, or both
* Provoked vulvodynia
* Unprovoked vulvodynia
* Women between 18 years of age and menopause

Exclusion Criteria:

* Pregnancy
* Menopause
* Interstitial cystitis
* Irritable bowel syndrome
* Untreated vaginitis
* Cervicitis
* Pelvic inflammatory disease
* Diagnosed with other pelvic pathology causing pain
* Concomitantly receiving physical therapy
* Concomitantly receiving biofeedback,
* Concomitantly receiving massage
* Concomitantly receiving additional acupuncture.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
vulvar pain | Baseline and 5 weeks
  Change from baseline in The Short Form McGill Pain Questionnaire at 5 weeks

SECONDARY OUTCOMES:
Dyspareunia | Baseline and 5 weeks
  Change from baseline in the pain subscale of the Female Sexual Function Index at 5 weeks

OTHER OUTCOMES:
Female sexual function | Baseline and 5 weeks
  Change from baseline in the total score of the Female Sexual Function Index at 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Schlaeger, PhD, Principal Investigator
Locations (1):
- Glenview Healing Arts, Glenview, Illinois, United States

REFERENCES:
- [Background] Stockdale CK, Lawson HW. 2013 Vulvodynia Guideline update. J Low Genit Tract Dis. 2014 Apr;18(2):93-100. doi: 10.1097/LGT.0000000000000021. PMID 24633161
- [Background] Curran S, Brotto LA, Fisher H, Knudson G, Cohen T. The ACTIV study: acupuncture treatment in provoked vestibulodynia. J Sex Med. 2010 Feb;7(2 Pt 2):981-95. doi: 10.1111/j.1743-6109.2009.01582.x. Epub 2009 Nov 12. PMID 19912491
- [Background] Danielsson I, Sjoberg I, Ostman C. Acupuncture for the treatment of vulvar vestibulitis: a pilot study. Acta Obstet Gynecol Scand. 2001 May;80(5):437-41. PMID 11328221
- [Background] Vickers AJ, Cronin AM, Maschino AC, Lewith G, MacPherson H, Foster NE, Sherman KJ, Witt CM, Linde K; Acupuncture Trialists' Collaboration. Acupuncture for chronic pain: individual patient data meta-analysis. Arch Intern Med. 2012 Oct 22;172(19):1444-53. doi: 10.1001/archinternmed.2012.3654. PMID 22965186